CLINICAL TRIAL: NCT04556760
Title: A Phase 2a Randomised, Double Blind, Multi-centre Study to Assess the Effect on Glucose Homeostasis of Two Dose Levels of AZD9567, Compared to Prednisolone, in Adults With Type 2 Diabetes
Brief Title: Study to Assess the Effect on Glucose Homeostasis of Two Dose Levels of AZD9567, Compared to Prednisolone, in Adults With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D6470C00005
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes Mellitus; Glucose Homeostasis; Pharmacodynamic; AZD9567; Prednisolone
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AZD9567; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both participants and investigators will be blinded. Investigators will remain blinded to each participant's assigned study intervention throughout the course of the study. In order to maintain this blind, a third party will be responsible for the reconstitution and dispensation of all study interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants will be randomised in a ratio of 1:1 to receive AZD9567 and prednisolone over two 72 hour periods in a cross over design (72 mg AZD9567 followed by 40 mg prednisolone [AB sequence group] or 40 mg prednisolone followed by 72 mg AZD9567 [BA sequence group]).
  Interventions: Drug: AZD9567; Drug: Prednisolone
- Cohort 2 (Experimental): Participants will be randomised in a ratio of 1:1 to receive AZD9567 and prednisolone over two 72 hour periods in a cross over design (40 mg AZD9567 followed by 20 mg prednisolone [AB sequence group] or 20 mg prednisolone followed by 40 mg AZD9567 [BA sequence group]).
  Interventions: Drug: AZD9567; Drug: Prednisolone
- Cohort 3 (Active Comparator): Participants will be randomised in a ratio of 1:1 to receive placebo and prednisolone over two 72 hour periods in a cross over design (placebo followed by 5 mg prednisolone [AB sequence group] or 5 mg prednisolone followed by placebo [BA sequence group]).
  Interventions: Drug: Prednisolone; Other: Placebo

INTERVENTIONS:
Drug: AZD9567 — Participants will receive 72 mg/day (oral suspension) of AZD9567 for 3 consecutive days of each treatment period in Cohort 1 and 40 mg/day for 3 consecutive days of each treatment period in Cohort 2.
  Arms: Cohort 1; Cohort 2
Drug: Prednisolone — Participants will receive 40 mg/day of prednisolone for 3 consecutive days of each treatment period in Cohort 1, 20 mg/day of prednisolone for 3 consecutive days of each treatment period in Cohort 2, and 5 mg/day prednisolone for 3 consecutive days of each treatment period in Cohort 3.
Other: Placebo — Participants will receive placebo for 3 consecutive days of each treatment period in Cohort 3.
  Arms: Cohort 3

SUMMARY:
The study is intended to assess the effect on glycaemic control of AZD9567, as measured by the glucose AUC(0-4) versus baseline following a standardised mixed meal tolerance test (MMTT), compared to prednisolone in adults with type 2 diabetes mellitus (T2DM). The study will also evaluate the safety, tolerability, and pharmacokinetics (PK) of AZD9567.

DETAILED DESCRIPTION:
This is a randomised, double blind, multi-centre, double dummy, and two-way cross-over study.

There will be a total of three cohorts. Each cohort will be treated for two 72-hour periods in a cross-over design, with a 3-week washout period between treatment periods. The total length of participant engagement (from screening to follow-up) is 79 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants with diagnosis of T2DM for 6 months prior to screening: HbA1c in the diabetes range or fasting plasma glucose 126 -220 mg/dL.
* On stable metformin therapy for at least 4 weeks, where no significant dose change (increase or decrease ≥ 500 mg/day) has occurred prior to screening and HbA1c 6% - 9.5%, or on dual therapy with metformin in combination with SGLT2i or DPP4i and HbA1c 6% - 8%. Participants on dual therapy will require 2 weeks wash-out of SGLT2i or DPP4i.
* Venous access suitable for multiple cannulations
* Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Female participants must be not lactating and not of childbearing potential.
* If sexually active, nonsterilized males who have a female partner of childbearing potential must practice effective contraceptive measures.
* Capable of giving signed informed consent.
* Provision of informed consent prior to any study specific procedures.

Exclusion Criteria:

* History or presence of type 1 diabetes.
* History of severe hypoglycaemia or hypoglycaemia unawareness within the last 6 months.
* History or presence of diabetic foot ulcers
* Participants with advanced diabetic complications.
* History of clinically significant lactic acidosis or ketoacidosis following diagnosis with T2DM.
* History of, or known significant infection or positivity at Visit 1, including hepatitis A, B, or C, HIV, tuberculosis that may put the participant at risk during participation in the study.
* History and / or presence of COVID-19.
* Donation of blood (≥ 450 mL) within 3 months or donation of plasma within 14 days before Visit 1.
* History of or current alcohol or drug abuse (including marijuana), as judged by the investigator.
* Previous psychiatric disorders.
* Any latent, acute, or chronic infections or at risk of infection, or history of skin abscesses within 90 days prior to the first administration of investigational medicinal product (IMP) at the discretion of the investigator.
* History of adrenal insufficiency.
* History or current inflammatory disorder.
* Any other condition that, in the opinion of the investigator, would interfere with evaluations of the IMP or interpretation of participant safety or study results.
* History of severe allergy/hypersensitivity to AZD9567 or any of the excipients of the product, or ongoing clinically important allergy/hypersensitivity as judged by the investigator.
* Oral or parenteral steroids 8 weeks prior to randomisation and during the study. Topical and inhaled steroids 4 weeks prior to randomisation are acceptable.
* Use of any prohibited medication during the study or if the required washout time of such medication was not adhered to.
* Receipt of live or live attenuated vaccine within 4 weeks prior to the first administration of IMP.
* Planned in-patient surgery, major dental procedure, or hospitalisation during the study.
* Previous participation or participation in any other research study within 1 month prior to Visit 1.
* Patient treated with any investigational drug within 30 days (or 5 half-lives, whichever is longer) prior to Visit 1.
* Uncontrolled hypertension (BP > 160 mmHg systolic or > 95 mmHg diastolic).
* Diagnosis of heart failure and current symptoms regardless of definition, ie, HfpEF, HfrEF.
* Acute coronary syndrome / unstable angina, coronary intervention procedures (percutaneous coronary intervention or coronary artery bypass graft) within the past 6 months.
* Stroke within the past 3 months.
* QTcF > 470 ms or family history of long QT-syndrome.
* AV-block II-III or sinus node dysfunction with significant pause, not treated with pacemaker.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, Principal Investigator — Profil Institut fur Stoffwechselforschung GmbH
Locations (3):
- Germany (3):
  - Research Site, Mainz
  - Research Site, Mannheim
  - Research Site, Neuss

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
  Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6470C00005&attachmentIdentifier=d1a10878-6b4a-4320-a661-b3f7986b52b2&fileName=AZ_COMPASS_D6470C00005_(PXL_248030)_Final_Draft_SAP_Redacted.pdf&versionIdentifier=
- See also: Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6470C00005&attachmentIdentifier=f2221f84-9958-4ffd-8e89-e2f6ca7a105e&fileName=AZ_COMPASS_D6470C00005_(PXL_248030)_Final_Draft_Protocol_Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6470C00005&attachmentIdentifier=5e02de02-bcd6-4401-ba0c-ae4becfb8118&fileName=AZ_COMPASS_D6470C00005_(PXL_248030)_Final_Draft_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in Germany between 26 November 2020 and 09 June 2021.
Pre-assignment Details: Patients with type 2 diabetes mellitus who met all the eligibility criteria were randomised in a ratio of 1:1 to a cohort and sequence group. Each cohort was treated for two 72 hour periods in a cross-over design, with a 3-week washout period between treatment periods.
Groups:
- Cohort 1: 72 mg AZD9567 First, Then 40 mg Prednisolone: Patients were randomised in a ratio of 1:1 to receive 72 mg AZD9567 followed by 40 mg prednisolone
- Cohort 1:40 mg Prednisolone First, Then 72 mg AZD9567: Patients were randomised in a ratio of 1:1 to receive 40 mg prednisolone followed by 72 mg AZD9567
- Cohort 2: 40 mg AZD9567 First, Then 20 mg Prednisolone: Patients were randomised in a ratio of 1:1 to receive 40 mg AZD9567 followed by 20 mg prednisolone
- Cohort 2: 20mg Prednisolone First, Then 40 mg AZD9567: Patients were randomised in a ratio of 1:1 to receive 20 mg prednisolone followed by 40 mg AZD9567
- Cohort 3: Placebo First, Then 5 mg Prednisolone: Patients were randomised in a ratio of 1:1 to receive placebo followed by 5 mg prednisolone
- Cohort 3: 5 mg Prednisolone First, Then Placebo: Patients were randomised in a ratio of 1:1 to receive 5 mg prednisolone followed by placebo
Period: Treatment Period 1 (72 Hours)
Arm/Group | Cohort 1: 72 mg AZD9567 First, Then 40 mg Prednisolone | Cohort 1:40 mg Prednisolone First, Then 72 mg AZD9567 | Cohort 2: 40 mg AZD9567 First, Then 20 mg Prednisolone | Cohort 2: 20mg Prednisolone First, Then 40 mg AZD9567 | Cohort 3: Placebo First, Then 5 mg Prednisolone | Cohort 3: 5 mg Prednisolone First, Then Placebo
Started | 14 | 14 | 5 | 4 | 4 | 5
Completed | 14 | 13 | 5 | 3 | 4 | 5
Not Completed | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Positive SARS-CoV-2 rapid test for patient's daughter | 0 | 0 | 0 | 1 | 0 | 0
Period: Washout Period (3 Weeks)
Arm/Group | Cohort 1: 72 mg AZD9567 First, Then 40 mg Prednisolone | Cohort 1:40 mg Prednisolone First, Then 72 mg AZD9567 | Cohort 2: 40 mg AZD9567 First, Then 20 mg Prednisolone | Cohort 2: 20mg Prednisolone First, Then 40 mg AZD9567 | Cohort 3: Placebo First, Then 5 mg Prednisolone | Cohort 3: 5 mg Prednisolone First, Then Placebo
Started | 14 | 13 | 5 | 3 | 4 | 5
Completed | 14 | 13 | 5 | 3 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (72 Hours)
Arm/Group | Cohort 1: 72 mg AZD9567 First, Then 40 mg Prednisolone | Cohort 1:40 mg Prednisolone First, Then 72 mg AZD9567 | Cohort 2: 40 mg AZD9567 First, Then 20 mg Prednisolone | Cohort 2: 20mg Prednisolone First, Then 40 mg AZD9567 | Cohort 3: Placebo First, Then 5 mg Prednisolone | Cohort 3: 5 mg Prednisolone First, Then Placebo
Started | 14 | 13 | 5 | 3 | 4 | 5
Completed | 14 | 13 | 5 | 3 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) consisted of all randomised patients who received at least 1 dose of study treatment.
Groups:
- Cohort 1: Patients were randomised in a ratio of 1:1 to receive 72 mg AZD9567 followed by 40 mg prednisolone or 40 mg prednisolone followed by 72 mg AZD9567
- Cohort 2: Patients were randomised in a ratio of 1:1 to receive 40 mg AZD9567 followed by 20 mg prednisolone or 20 mg prednisolone followed by 40 mg AZD9567
- Cohort 3: Patients were randomised in a ratio of 1:1 to receive placebo followed by 5 mg prednisolone or 5 mg prednisolone followed by placebo
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 27 | 8 | 9 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.3 (6.41) | 64.4 (9.32) | 66.6 (5.36) | 66.6 (6.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 1 | 7
  Male | 23 | 6 | 8 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 8 | 9 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 26 | 7 | 9 | 42
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glucose Area Under the Plasma Concentration Versus Time Curve From Zero to 4 Hours Post-dose AUC(0-4)
Description: The change from baseline in glucose AUC(0-4) was analysed to determine the Pharmacodynamic (PD) effect of AZD9567 compared to Prednisolone following a standardised Mixed meal tolerance test (MMTT).
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Days -1 (baseline), and Days 4 (Treatment period 1 and 2)
Population: Full Analysis Set (FAS) consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: minute*millimole/liter (min*mmol/L)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
minute*millimole/liter (min*mmol/L)
  AZD9567: number analyzed (Participants) | 27 | 8 | 0
  AZD9567 | -190.0296 (63.8805) | -182.7172 (149.8600) |
  Prednisolone | -57.0768 (63.8762) | -40.6842 (141.7154) | -184.9677 (88.9807)
  Placebo: number analyzed (Participants) | 0 | 0 | 9
  Placebo |  |  | -311.8506 (88.5443)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg); Test type: Other; p = 0.036, Mixed Models Analysis; Mean Difference (Final Values) = -132.9528, 95% CI 2-sided [-256.5082 to -9.3973]
Statistical Analysis 2: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg); Test type: Other; p = 0.432, Mixed Models Analysis; Mean Difference (Final Values) = -142.0330, 95% CI 2-sided [-554.8722 to 270.8061]
Statistical Analysis 3: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5mg); Test type: Other; p = 0.030, Mixed Models Analysis; Mean Difference (Final Values) = -126.8829, 95% CI 2-sided [-236.0426 to -17.7233]

2. Secondary Outcome: Mean Glucose Level as Determined Via the Continuous Glucose Monitoring (CGM) System
Description: The mean glucose levels in mmol/L at 48-72 h was analysed to determine the effect of AZD9567 on CGM compared to prednisolone.
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: 48 to 72 hours
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: millimole/liter (mmol/L) per day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
millimole/liter (mmol/L) per day
  AZD9567: number analyzed (Participants) | 27 | 8 | 0
  AZD9567 | 8.5730 (0.3114) | 7.7870 (0.2517) |
  Prednisolone: number analyzed (Participants) | 26 | 8 | 9
  Prednisolone | 10.0797 (0.3150) | 8.8969 (0.2494) | 7.4238 (0.2889)
  Placebo: number analyzed (Participants) | 0 | 0 | 9
  Placebo |  |  | 7.2638 (0.2888)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg); Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.5067, 95% CI 2-sided [-2.0820 to -0.9314]
Statistical Analysis 2: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg); Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.1099, 95% CI 2-sided [-1.7257 to -0.4941]
Statistical Analysis 3: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5mg); Test type: Other; p = 0.547, Mixed Models Analysis; Mean Difference (Final Values) = -0.1601, 95% CI [-0.6930 to 0.3729]

3. Secondary Outcome: Rise in Mean Glucose Levels Over 24-hour Periods From Start of IMP Dosing
Description: The mean glucose level in mmol/L was analysed to determine the effect of AZD9567 on CGM compared to prednisolone.
  For the calculation of the rise in mean glucose levels, the baseline was the average of the values from -24 hours to first dosing on Day 1 of each period.
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: Baseline and up to 72 hours (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L per day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
mmol/L per day
  AZD9567 (00 to 24 hours [h]): number analyzed (Participants) | 27 | 8 | 0
  AZD9567 (00 to 24 hours [h]) | 1.2071 (0.2869) | 0.4070 (0.2509) |
  Prednisolone (00 to 24 h): number analyzed (Participants) | 26 | 8 | 9
  Prednisolone (00 to 24 h) | 2.7086 (0.2938) | 1.2545 (0.2460) | 0.3123 (0.1549)
  Placebo (00 to 24 h): number analyzed (Participants) | 0 | 0 | 9
  Placebo (00 to 24 h) |  |  | -0.0477 (0.1547)
  AZD9567 (24 to 48 h): number analyzed (Participants) | 27 | 8 | 0
  AZD9567 (24 to 48 h) | 0.8011 (0.2978) | 0.5428 (0.2483) |
  Prednisolone (24 to 48 h): number analyzed (Participants) | 26 | 8 | 9
  Prednisolone (24 to 48 h) | 2.6653 (0.3044) | 1.3206 (0.2448) | -0.2415 (0.2898)
  Placebo (24 to 48 h): number analyzed (Participants) | 0 | 0 | 9
  Placebo (24 to 48 h) |  |  | -0.3260 (0.2894)
  AZD9567 (48 to 72 h): number analyzed (Participants) | 27 | 8 | 0
  AZD9567 (48 to 72 h) | 0.8529 (0.3210) | 0.0744 (0.2714) |
  Prednisolone (48 to 72 h): number analyzed (Participants) | 26 | 8 | 9
  Prednisolone (48 to 72 h) | 2.4527 (0.3274) | 1.2174 (0.2664) | -0.2202 (0.2229)
  Placebo (48 to 72 h): number analyzed (Participants) | 0 | 0 | 9
  Placebo (48 to 72 h) |  |  | -0.3500 (0.2224)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg [00 to 24 h]); Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.5015, 95% CI 2-sided [-2.2258 to -0.7773]
Statistical Analysis 2: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg [24 to 48 h]); Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.8643, 95% CI [-2.5611 to -1.1674]
Statistical Analysis 3: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg [48 to 72 h]); Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.5998, 95% CI 2-sided [-2.3025 to -0.8971]
Statistical Analysis 4: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg [00 to 24 h]); Test type: Other; p = 0.013, Mixed Models Analysis; Mean Difference (Final Values) = -0.8474, 95% CI 2-sided [-1.4465 to -0.2484]
Statistical Analysis 5: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg [24 to 48 h]); Test type: Other; p = 0.061, Mixed Models Analysis; Mean Difference (Final Values) = -0.7778, 95% CI 2-sided [-1.6022 to 0.0466]
Statistical Analysis 6: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg [48 to 72 h]); Test type: Other; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -1.1430, 95% CI 2-sided [-1.7622 to -0.5238]
Statistical Analysis 7: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5 mg [00 to 24 h]); Test type: Other; p = 0.125, Mixed Models Analysis; Mean Difference (Final Values) = -0.3600, 95% CI 2-sided [-0.8338 to 0.1138]
Statistical Analysis 8: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5 mg [24 to 48 h]); Test type: Other; p = 0.840, Mixed Models Analysis; Mean Difference (Final Values) = -0.0845, 95% CI 2-sided [-0.9706 to 0.8016]
Statistical Analysis 9: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5 mg [48 to 72 h]); Test type: Other; p = 0.571, Mixed Models Analysis; Mean Difference (Final Values) = -0.1298, 95% CI 2-sided [-0.6460 to 0.3864]

4. Secondary Outcome: Change From Baseline in Fasting Glucose
Description: Pharmacodynamic effects (fasting glucose) of AZD9567 following a MMTT were evaluated as compared to prednisolone.
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Day -1 (Baseline), and Day 4 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
mmol/L
  AZD9567: number analyzed (Participants) | 27 | 8 | 0
  AZD9567 | -1.14 (0.17) | -0.95 (0.36) |
  Prednisolone | -1.06 (0.17) | -0.91 (0.35) | -1.15 (0.20)
  Placebo: number analyzed (Participants) | 0 | 0 | 9
  Placebo |  |  | -1.15 (0.20)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg); Test type: Other; p = 0.753, Mixed Models Analysis; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.55 to 0.40]
Statistical Analysis 2: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg); Test type: Other; p = 0.802, Mixed Models Analysis; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.46 to 0.37]
Statistical Analysis 3: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5mg); Test type: Other; p = 0.985, Mixed Models Analysis; Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.37 to 0.37]

5. Secondary Outcome: Change From Baseline AUC(0-4) on Hormones Related to Glucose Homeostasis (Insulin)
Description: Effects of AZD9567 on insulin AUC(0-4) were assessed following MMTT compared to prednisolone.
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Day -1 (Baseline), and Day 4 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: minute*picomole/liter (min*pmole/L)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
minute*picomole/liter (min*pmole/L)
  AZD9567: number analyzed (Participants) | 21 | 8 | 0
  AZD9567 | 15319.3857 (4165.9135) | 13413.1929 (4791.9873) |
  Prednisolone: number analyzed (Participants) | 23 | 7 | 9
  Prednisolone | -5179.3659 (3989.2683) | 10091.7869 (5461.2631) | 4915.4115 (7049.5460)
  Placebo: number analyzed (Participants) | 0 | 0 | 9
  Placebo |  |  | 2216.5532 (7049.0432)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg); Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 20498.7, 95% CI 2-sided [10819.2 to 30178.2]
Statistical Analysis 2: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg); Test type: Other; p = 0.659, Mixed Models Analysis; Mean Difference (Final Values) = 3321.4, 95% CI 2-sided [-12975.8 to 19618.6]
Statistical Analysis 3: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5mg); Test type: Other; p = 0.521, Mixed Models Analysis; Mean Difference (Final Values) = -2698.8, 95% CI 2-sided [-14849.0 to 9451.3]

6. Secondary Outcome: Change From Baseline AUC(0-4) on Hormones Related to Glucose Homeostasis (Glucagon)
Description: Effects of AZD9567 on glucagon AUC(0-4) were assessed following MMTT in comparison to prednisolone.
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Day -1 (Baseline), and Day 4 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: min*pmol/L
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
min*pmol/L
  AZD9567: number analyzed (Participants) | 27 | 8 | 0
  AZD9567 | -36.9846 (216.5777) | 552.0634 (213.9300) |
  Prednisolone | 965.6018 (216.6054) | 511.0798 (213.5970) | 259.9835 (298.9801)
  Placebo: number analyzed (Participants) | 0 | 0 | 7
  Placebo |  |  | 361.3971 (348.5104)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg); Test type: Other; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -1002.5864, 95% CI 2-sided [-1620.2150 to -384.9577]
Statistical Analysis 2: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg); Test type: Other; p = 0.865, Mixed Models Analysis; Mean Difference (Final Values) = 40.9836, 95% CI 2-sided [-526.6968 to 608.6640]
Statistical Analysis 3: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5mg); Test type: Other; p = 0.754, Mixed Models Analysis; Mean Difference (Final Values) = 101.4137, 95% CI 2-sided [-628.8097 to 831.6370]

7. Secondary Outcome: Change From Baseline AUC(0-4) on Hormones Related to Glucose Homeostasis (Glucagon-like Peptide-1 [GLP-1])
Description: Effects of AZD9567 on GLP-1 AUC(0-4) were assessed following MMTT in comparison to prednisolone.
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Day -1 (Baseline), and Day 4 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: min*pmol/L
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
min*pmol/L
  AZD9567: number analyzed (Participants) | 27 | 8 | 0
  AZD9567 | 615.9803 (328.8418) | 322.5690 (454.2028) |
  Prednisolone | 1841.8853 (328.8877) | 789.5492 (450.2548) | 575.6726 (318.1088)
  Placebo: number analyzed (Participants) | 0 | 0 | 9
  Placebo |  |  | 200.3565 (317.6326)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg); Test type: Other; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = -1225.9050, 95% CI 2-sided [-2007.2241 to -444.5859]
Statistical Analysis 2: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg); Test type: Other; p = 0.313, Mixed Models Analysis; Mean Difference (Final Values) = -466.9802, 95% CI 2-sided [-1521.5088 to 587.5485]
Statistical Analysis 3: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5mg); Test type: Other; p = 0.404, Mixed Models Analysis; Mean Difference (Final Values) = -375.3161, 95% CI [-1433.6265 to 682.9943]

8. Secondary Outcome: Change From Baseline AUC(0-4) on Hormones Related to Glucose Homeostasis (Glucose-dependent Insulin Releasing Polypeptide [GIP])
Description: Effects of AZD9567 on GIP AUC(0-4) were assessed following MMTT in comparison to prednisolone.
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Day -1 (Baseline), and Day 4 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: min*pmol/L
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
min*pmol/L
  AZD9567: number analyzed (Participants) | 27 | 8 | 0
  AZD9567 | 3658.9885 (584.5079) | 3842.9307 (1303.1553) |
  Prednisolone: number analyzed (Participants) | 26 | 8 | 9
  Prednisolone | 3293.3563 (596.7472) | 3654.6947 (1289.5516) | 3271.5164 (823.9967)
  Placebo: number analyzed (Participants) | 0 | 0 | 9
  Placebo |  |  | 2210.0670 (827.7335)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg); Test type: Other; p = 0.608, Mixed Models Analysis; Mean Difference (Final Values) = 365.6323, 95% CI 2-sided [-1097.7973 to 1829.0618]
Statistical Analysis 2: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg); Test type: Other; p = 0.897, Mixed Models Analysis; Mean Difference (Final Values) = 188.2360, 95% CI 2-sided [-3214.3323 to 3590.8043]
Statistical Analysis 3: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5mg); Test type: Other; p = 0.381, Mixed Models Analysis; Mean Difference (Final Values) = -1061.4494, 95% CI [-3588.2233 to 1465.3244]

9. Secondary Outcome: Change From Baseline in AUC(0-4) on C-peptide
Description: Effects of AZD9567 on C-peptide AUC(0-4) were assessed through a MMTT in comparison to prednisolone.
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Day -1 (Baseline), and Day 4 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: minute*nanomole/L (min*nmol/L)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
minute*nanomole/L (min*nmol/L)
  AZD9567: number analyzed (Participants) | 27 | 8 | 0
  AZD9567 | 85.3305 (13.4279) | 82.1134 (22.9858) |
  Prednisolone | 24.9094 (13.4282) | 55.6606 (22.6155) | 24.7245 (22.2183)
  Placebo: number analyzed (Participants) | 0 | 0 | 9
  Placebo |  |  | 0.7002 (22.0424)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg); Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 60.4211, 95% CI [29.4904 to 91.3518]
Statistical Analysis 2: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg); Test type: Other; p = 0.432, Mixed Models Analysis; Mean Difference (Final Values) = 26.4529, 95% CI [-44.9414 to 97.8471]
Statistical Analysis 3: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5mg); Test type: Other; p = 0.282, Mixed Models Analysis; Mean Difference (Final Values) = -24.0243, 95% CI [-74.0731 to 26.0245]

10. Secondary Outcome: Change From Baseline in Ratio of Insulin to Glucose Level Between 10 and 0 Minutes (ΔI10/ΔG10)
Description: Effects of AZD9567 on ΔI10/ΔG10 of beta cell function from the MMTT compared to Prednisolone was evaluated.
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Day -1 (Baseline), and Day 4 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
Ratio
  AZD9567: number analyzed (Participants) | 16 | 8 | 0
  AZD9567 | -0.5249 (0.6632) | NA (NA) — Convergence was not met thus no data are available. |
  Prednisolone: number analyzed (Participants) | 18 | 8 | 5
  Prednisolone | 0.0774 (0.6674) | NA (NA) — Convergence was not met thus no data are available. | -0.8153 (0.8305)
  Placebo: number analyzed (Participants) | 0 | 0 | 7
  Placebo |  |  | -0.3532 (0.6893)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg); Test type: Other; p = 0.531, Mixed Models Analysis; Mean Difference (Final Values) = -0.6023, 95% CI 2-sided [-2.5463 to 1.3416]
Statistical Analysis 2: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5mg); Test type: Other; p = 0.682, Mixed Models Analysis; Mean Difference (Final Values) = 0.4621, 95% CI 2-sided [-2.0933 to 3.0176]

11. Secondary Outcome: Change From Baseline in Ratio of Insulin to Glucose Level Between 30 and 0 Minutes [ΔI30/ΔG30])
Description: Effects of AZD9567 on ΔI30/ΔG30 of beta cell function from the MMTT compared to Prednisolone was evaluated.
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Day -1 (Baseline), and Day 4 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
Ratio
  AZD9567: number analyzed (Participants) | 25 | 8 | 0
  AZD9567 | 0.1203 (0.0726) | 0.1824 (0.0773) |
  Prednisolone: number analyzed (Participants) | 24 | 6 | 8
  Prednisolone | 0.0530 (0.0755) | 0.0943 (0.1264) | -0.1047 (0.0665)
  Placebo: number analyzed (Participants) | 0 | 0 | 9
  Placebo |  |  | 0.0209 (0.0599)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg); Test type: Other; p = 0.526, Mixed Models Analysis; Mean Difference (Final Values) = 0.0679, 95% CI [-0.1520 to 0.2866]
Statistical Analysis 2: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg; Test type: Other; p = 0.569, Mixed Models Analysis; Mean Difference (Final Values) = 0.0882, 95% CI [-0.2653 to 0.4416]
Statistical Analysis 3: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5mg); Test type: Other; p = 0.166, Mixed Models Analysis; Mean Difference (Final Values) = 0.1257, 95% CI 2-sided [-0.0677 to 0.3191]

12. Secondary Outcome: Change From Baseline in Ratio of C-peptide to Glucose Level Between 10 and 0 Minutes (ΔC10/ΔG10)
Description: Effects of AZD9567 on ΔC10/ΔG10 of beta cell function from the MMTT compared to Prednisolone was evaluated.
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Day -1 (Baseline), and Day 4 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
Ratio
  AZD9567: number analyzed (Participants) | 17 | 6 | 0
  AZD9567 | -0.0004 (0.0095) | 0.0059 (0.0041) |
  Prednisolone: number analyzed (Participants) | 20 | 4 | 6
  Prednisolone | -0.0103 (0.0092) | 0.0026 (0.0047) | -0.0033 (0.0064)
  Placebo: number analyzed (Participants) | 0 | 0 | 7
  Placebo |  |  | -0.0024 (0.0057)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg); Test type: Other; p = 0.226, Mixed Models Analysis; Mean Difference (Final Values) = 0.0100, 95% CI 2-sided [-0.0072 to 0.0271]
Statistical Analysis 2: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg); Test type: Other; p = 0.619, Mixed Models Analysis; Mean Difference (Final Values) = 0.0033, 95% CI [-0.0128 to 0.0195]
Statistical Analysis 3: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5mg); Test type: Other; p = 0.917, Mixed Models Analysis; Mean Difference (Final Values) = 0.0009, 95% CI [-0.0189 to 0.0207]

13. Secondary Outcome: Change From Baseline in Ratio of C-peptide to Glucose Level Between 30 and 0 Minutes (ΔC30/ΔG30)
Description: Effects of AZD9567 on ΔC30/ΔG30 of beta cell function from the MMTT compared to Prednisolone was evaluated.
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Day -1 (Baseline), and Day 4 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
Ratio
  AZD9567: number analyzed (Participants) | 27 | 8 | 0
  AZD9567 | 0.0012 (0.0005) | 0.0007 (0.0005) |
  Prednisolone | 0.0005 (0.0005) | 0.0004 (0.0005) | -0.0010 (0.0005)
  Placebo: number analyzed (Participants) | 0 | 0 | 9
  Placebo |  |  | 0.0002 (0.0005)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg); Test type: Other; p = 0.357, Mixed Models Analysis; Mean Difference (Final Values) = 0.0007, 95% CI 2-sided [-0.0008 to 0.0022]
Statistical Analysis 2: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg); Test type: Other; p = 0.676, Mixed Models Analysis; Mean Difference (Final Values) = 0.0003, 95% CI 2-sided [-0.0012 to 0.0017]
Statistical Analysis 3: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5mg); Test type: Other; p = 0.096, Mixed Models Analysis; Mean Difference (Final Values) = 0.0012, 95% CI [-0.0002 to 0.0026]

14. Secondary Outcome: Change From Baseline in 24-hour Urinary Potassium Excretion
Description: The concentration of potassium in urine was measured over 24 hours to determine the effect of AZD9567 on urinary potassium (U-K) excretion compared to prednisolone.
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Day -1 (Baseline), and Day 4 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: mmol/day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
mmol/day
  AZD9567: number analyzed (Participants) | 27 | 8 | 0
  AZD9567 | -2.92 (3.27) | -6.05 (4.30) |
  Prednisolone | -1.19 (3.27) | 4.92 (4.29) | -2.49 (9.08)
  Placebo: number analyzed (Participants) | 0 | 0 | 9
  Placebo |  |  | -2.85 (9.07)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg); Test type: Other; p = 0.646, Mixed Models Analysis; Mean Difference (Final Values) = -1.73, 95% CI 2-sided [-9.40 to 5.95]
Statistical Analysis 2: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg); Test type: Other; p = 0.110, Mixed Models Analysis; Mean Difference (Final Values) = -10.97, 95% CI [-25.39 to 3.44]
Statistical Analysis 3: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5mg); Test type: Other; p = 0.932, Mixed Models Analysis; Mean Difference (Final Values) = -0.35, 95% CI [-10.32 to 9.61]

15. Secondary Outcome: Change From Baseline in 24-hour Urinary Sodium Excretion
Description: The concentration of sodium in urine was measured over 24 hours to determine the effect of AZD9567 on urinary-sodium (U-Na) excretion compared to prednisolone.
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Day -1 (Baseline), and Day 4 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: mmol/day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
mmol/day
  AZD9567: number analyzed (Participants) | 27 | 8 | 0
  AZD9567 | 17.4 (11.0) | 39.9 (20.4) |
  Prednisolone | 9.7 (11.0) | 17.6 (20.3) | -18.1 (21.4)
  Placebo: number analyzed (Participants) | 0 | 0 | 9
  Placebo |  |  | 12.9 (21.3)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg); Test type: Other; p = 0.533, Mixed Models Analysis; Mean Difference (Final Values) = 7.6, 95% CI 2-sided [-17.4 to 32.7]
Statistical Analysis 2: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg); Test type: Other; p = 0.311, Mixed Models Analysis; Mean Difference (Final Values) = 22.3, 95% CI [-26.7 to 71.3]
Statistical Analysis 3: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5mg); Test type: Other; p = 0.204, Mixed Models Analysis; Mean Difference (Final Values) = 31.0, 95% CI [-21.9 to 83.9]

16. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Zero to the Last Quantifiable Concentration (AUClast)
Description: AUClast of AZD9567 following once daily dosing was evaluated.
Time Frame: Upto 30 hours post dose (Treatment period 1 and 2)
Population: Pharmacokinetic analysis set (PKAS) consisted of all patients in the FAS with at least 1 quantifiable AZD9567 concentration and no important protocol deviations, or adverse events (AEs) considered to have an effect upon PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanomole/liter (h*nmol/L)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 8
hour*nanomole/liter (h*nmol/L) | 34400 (42.97) | 18410 (46.06)

17. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Zero to 24 Hours Post-dose [AUC(0-24)]
Description: AUC(0-24) of AZD9567 following once daily dosing was evaluated.
Time Frame: 24 hours post dose
Population: PKAS consisted of all patients in the FAS with at least 1 quantifiable AZD9567 concentration and no important protocol deviations, or AEs considered to have an effect upon PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 8
h*nmol/L | 32920 (41.32) | 17790 (44.86)

18. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Zero to 6 Hours Post-dose [AUC(0-6)]
Description: AUC(0-6) of AZD9567 following once daily dosing was evaluated.
Time Frame: 6 hours post dose
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 8
h*nmol/L | 17050 (30.45) | 9914 (35.06)

19. Secondary Outcome: Maximum Observed Drug Concentration (Cmax)
Description: Cmax of AZD9567 following once daily dosing was evaluated.
Time Frame: Upto 30 hours post dose (Treatment period 1 and 2)
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 8
nmol/L | 4501 (26.90) | 2939 (31.50)

20. Secondary Outcome: Time to Reach Maximum Observed Drug Concentration (Tmax)
Description: Tmax of AZD9567 following once daily dosing was evaluated.
Time Frame: Upto 30 hours post dose (Treatment period 1 and 2)
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 8
hours | 0.50 [0.25 to 1.50] | 0.50 [0.50 to 1.00]

21. Secondary Outcome: Terminal Elimination Half-life (t½λz)
Description: t½λz of AZD9567 following once daily dosing was evaluated.
Time Frame: Upto 30 hours post dose (Treatment period 1 and 2)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 8
hours | 6.99 (1.44) | 6.16 (1.08)

22. Secondary Outcome: Apparent Total Body Clearance of Drug From Plasma After Extravascular (CL/F)
Description: CL/F of AZD9567 following once daily dosing was evaluated.
Time Frame: Upto 30 hours post dose (Treatment period 1 and 2)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Liter/hour (L/h)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 8
Liter/hour (L/h) | 4.766 (1.896) | 4.924 (2.098)

23. Secondary Outcome: Apparent Volume of Distribution Following Extravascular Administration (Vz/F)
Description: Vz/F of AZD9567 was derived using standard non-compartmental methods using WinNonLin version 8.1 or higher (Certara).
Time Frame: Upto 30 hours post dose (Treatment period 1 and 2)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 8
Liter | 45.11 (11.39) | 41.75 (14.19)

24. Secondary Outcome: Tumour Necrosis Factor Alpha (TNFα) Concentrations
Description: Relationship between AZD9567 exposure and inhibition of LPS-stimulated TNFα release for high and low dose comparison (Cohort 1 and Cohort 2) was assessed. LPS-stimulated TNFα concentration was measured.
Time Frame: On Days 3 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: nanogram/liter (ng/L)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 27 | 8
nanogram/liter (ng/L)
  AZD9567 (0h): number analyzed (Participants) | 26 | 8
  AZD9567 (0h) | 21000.1 (15413.92) | 23525.0 (15260.57)
  Prednisolone (0h): number analyzed (Participants) | 26 | 8
  Prednisolone (0h) | 21361.5 (18124.60) | 12385.0 (11835.31)
  AZD9567 (1h): number analyzed (Participants) | 26 | 8
  AZD9567 (1h) | 9100.2 (6248.93) | 8122.5 (5303.16)
  Prednisolone (1h): number analyzed (Participants) | 25 | 8
  Prednisolone (1h) | 3581.1 (3642.93) | 3617.5 (1552.62)
  AZD9567 (2h): number analyzed (Participants) | 26 | 8
  AZD9567 (2h) | 8170.7 (5053.69) | 8098.0 (7709.06)
  Prednisolone (2h): number analyzed (Participants) | 26 | 8
  Prednisolone (2h) | 1648.2 (1109.64) | 1421.1 (591.80)
  AZD9567 (4h) | 7534.6 (4519.50) | 8898.8 (5249.73)
  Prednisolone (4h) | 2293.1 (1329.60) | 4292.0 (3207.76)
  AZD9567 (8h) | 10674.4 (7731.94) | 13023.8 (8946.33)
  Prednisolone (8h): number analyzed (Participants) | 26 | 8
  Prednisolone (8h) | 4585.7 (4453.61) | 7247.5 (2889.87)
  AZD9567 (12h) | 13332.5 (10831.44) | 14695.0 (11422.87)
  Prednisolone (12h) | 12415.5 (9474.44) | 16790.0 (8010.23)
  AZD9567 (24h) | 22136.7 (13414.45) | 19741.3 (11048.74)
  Prednisolone (24h) | 23292.9 (15548.12) | 20920.0 (14802.66)

25. Secondary Outcome: Change From Baseline AUC(0-4) on Hormones Related to Glucose Homeostasis (Free Fatty Acids)
Description: Effects of AZD9567 on free fatty acids were evaluated following a MMTT compared to prednisolone.
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Day -1 (Baseline), and Day 4 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: min*mmol/L
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
min*mmol/L
  AZD9567: number analyzed (Participants) | 27 | 8 | 0
  AZD9567 | -18.1304 (1.7543) | -14.0582 (3.7038) |
  Prednisolone | -14.1238 (1.7542) | -19.8117 (3.7060) | -4.1625 (3.7212)
  Placebo: number analyzed (Participants) | 0 | 0 | 9
  Placebo |  |  | 4.8995 (3.7153)
Statistical Analysis 1: Comparison: Cohort 1; Pairwise Comparisons with Prednisolone (AZD9567 72mg vs Prednisolone 40mg); Test type: Other; p = 0.103, Mixed Models Analysis; Mean Difference (Final Values) = -4.0066, 95% CI 2-sided [-8.8880 to 0.8748]
Statistical Analysis 2: Comparison: Cohort 2; Pairwise Comparisons with Prednisolone (AZD9567 40mg vs Prednisolone 20mg); Test type: Other; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = 5.7535, 95% CI [2.6034 to 8.9036]
Statistical Analysis 3: Comparison: Cohort 3; Pairwise Comparisons with Prednisolone (Placebo vs Prednisolone 5mg); Test type: Other; p = 0.023, Mixed Models Analysis; Mean Difference (Final Values) = 9.0619, 95% CI [1.6740 to 16.4499]

26. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment- Insulin Resistance (HOMA-IR)
Description: The HOMA-IR was calculated based on glucose and insulin measured prior to MMTT.
  HOMA-IR= Glucose(mmol/L) x Insulin (mU/L) / 22.5
  HOMA-IR score estimates the degree of insulin resistance. Higher range indicates greater insulin resistance (i.e. high diabetes risk), while lower range indicates insulin sensitivity (i.e. low diabetes risk)
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Day -1 (Baseline), and Day 4 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
Score
  AZD9567: number analyzed (Participants) | 26 | 8 | 0
  AZD9567 | -0.4406 (1.9875) | -0.1738 (0.7576) |
  Prednisolone: number analyzed (Participants) | 25 | 8 | 9
  Prednisolone | -0.7023 (1.5896) | 0.0721 (0.9606) | -0.5662 (0.7364)
  Placebo: number analyzed (Participants) | 0 | 0 | 9
  Placebo |  |  | -0.9280 (0.8173)

27. Secondary Outcome: Change From Baseline in HOMA-insulin Sensitivity (HOMA-S)
Description: Insulin sensitivity is a term used to indicate the responsiveness of the peripheral tissue cells to insulin, and their resultant capacity to uptake glucose out of the bloodstream.
  HOMA-S score estimates the degree of insulin sensitivity. HOMA-S was calculated as the reciprocal of HOMA-IR.
  Higher values indicates greater insulin sensitivity (i.e. low diabetes risk), while lower values indicates insulin resistance (i.e. high diabetes risk)
  In Cohort 1 and 2, Placebo was not administered, therefore in Placebo row the participants analyzed is kept as 0.
  In Cohort 3, AZD9567 was not administered, therefore in AZD9567 row the participants analyzed is kept 0.
Time Frame: On Day -1 (Baseline), and Day 4 (Treatment period 1 and 2)
Population: FAS consisted of all randomised patients who received at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 27 | 8 | 9
Score
  AZD9567: number analyzed (Participants) | 26 | 8 | 0
  AZD9567 | 0.0134 (0.2352) | -0.0360 (0.1990) |
  Prednisolone: number analyzed (Participants) | 25 | 8 | 9
  Prednisolone | 0.0328 (0.1400) | -0.0799 (0.2077) | 0.0750 (0.0949)
  Placebo: number analyzed (Participants) | 0 | 0 | 9
  Placebo |  |  | 0.1468 (0.0930)

28. Secondary Outcome: Number of Participants With Adverse Events
Description: Safety and tolerability of AZD9567 was assessed.
Time Frame: From screening up to 79 days
Population: Safety Analysis Set (SAF) consisted of all patients who were randomised to one of the 2 sequence groups within the cohort and have received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: AZD9567 72mg; Cohort 1: Prednisolone 40mg: Patients were randomised in a ratio of 1:1 to receive 72 mg AZD9567 followed by 40 mg prednisolone or 40 mg prednisolone followed by 72 mg AZD9567
- Cohort 2: AZD9567 40mg; Cohort 2: Prednisolone 20mg: Patients were randomised in a ratio of 1:1 to receive 40 mg AZD9567 followed by 20 mg prednisolone or 20 mg prednisolone followed by 40 mg AZD9567
- Cohort 3: Placebo; Cohort 3: Prednisolone 5mg: Patients were randomised in a ratio of 1:1 to receive placebo followed by 5 mg prednisolone or 5 mg prednisolone followed by placebo
Arm/Group | Cohort 1: AZD9567 72mg | Cohort 1: Prednisolone 40mg | Cohort 2: AZD9567 40mg | Cohort 2: Prednisolone 20mg | Cohort 3: Placebo | Cohort 3: Prednisolone 5mg
Number analyzed (Participants) | 27 | 27 | 8 | 8 | 9 | 9
Participants
  Any Adverse Event (AE) | 4 | 7 | 2 | 5 | 1 | 0
  Any AE with outcome = death | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE (including events with outcome = death) | 0 | 0 | 0 | 0 | 0 | 0
  Any AE leading to discontinuation of Investigational Product | 0 | 0 | 0 | 0 | 0 | 0
  Any AE leading to drug interruption | 0 | 0 | 0 | 0 | 0 | 0
  Any AE leading to withdrawal from study | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Screening up to Final/ end of treatment visit (Day 79).
Description: Safety Analysis Set (SAF) consisted of all patients who were randomised to one of the 2 sequence groups within the cohort and have received at least 1 dose of study intervention. The SAF was analysed according to actual treatment.
  Three additional arms were created to capture Adverse Events for each treatment within the cohort.
Groups:
- Cohort 1: AZD9567 72mg; Cohort 1: Prednisolone 40mg: Patients were randomised in a ratio of 1:1 to receive 72 mg AZD9567 followed by 40 mg prednisolone or 40 mg prednisolone followed by 72 mg AZD956
- Cohort 2: Prednisolone 20mg: Patients were randomised in a ratio of 1:1 to receive 40 mg AZD9567 followed by 20 mg prednisolone or 20 mg prednisolone followed by 40 mg AZD956
Arm/Group | Cohort 1: AZD9567 72mg | Cohort 1: Prednisolone 40mg | Cohort 2: AZD9567 40mg | Cohort 2: Prednisolone 20mg | Cohort 3: Placebo | Cohort 3: Prednisolone 5mg
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/8 | 0/8 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/8 | 0/8 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 4/27 | 7/27 | 2/8 | 5/8 | 1/9 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: AZD9567 72mg (N=27) | Cohort 1: Prednisolone 40mg (N=27) | Cohort 2: AZD9567 40mg (N=8) | Cohort 2: Prednisolone 20mg (N=8) | Cohort 3: Placebo (N=9) | Cohort 3: Prednisolone 5mg (N=9)
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 2 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Administration site phlebitis (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Catheter site erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information may be disclosed without prior written approval from AstraZeneca.

DOCUMENTS (2):
  • Study Protocol (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT04556760/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT04556760/SAP_001.pdf